CLINICAL TRIAL: NCT02467543
Title: The Efficacy of Viburnum Opulus 3X in the Treatment of Primary Dysmenorrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Johannesburg (Other)
Responsible Party: Principal Investigator, Dr J. Pellow, Dr Janice Pellow, University of Johannesburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZuleikaSaem200819247
Record Dates: First submitted 2015-06-05; First posted 2015-06-10 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Dysmenorrhea
Keywords: Primary dysmenorrhea; Viburnum opulus 3X; Homoeopathic
MeSH Terms: conditions — Dysmenorrhea | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 20% Ethanol (Placebo Comparator): 20% ethanol containing no active ingredients. Ten drops will be taken three times daily when the pain and cramping of dysmenorrhea start, and should be stopped when the pain and cramping have ceased.
  Interventions: Other: 20% Ethanol
- Viburnum opulus 3X (Experimental): Viburnum opulus 3X in a vehicle of 20% ethanol. Ten drops will be taken three times daily when the pain and cramping of dysmenorrhea start, and should be stopped when the pain and cramping have ceased.
  Interventions: Other: Viburnum opulus 3X

INTERVENTIONS:
Other: 20% Ethanol — Unmedicated 20% Ethanol
  Arms: 20% Ethanol
Other: Viburnum opulus 3X — Viburnum opulus 3X in a vehicle of 20% ethanol.
  Arms: Viburnum opulus 3X

SUMMARY:
Dysmenorrhea (painful menstruation) is a common gynaecological disorder that is prevalent in more than 50% of women during their reproductive years. Primary dysmenorrhea describes cyclic uterine pain without any identifiable or underlying causes. Menstrual pain results as a consequence of endometrial ischemia, high levels of prostaglandins and other inflammatory mediators. Conventional treatment for primary dysmenorrhea consists of non-steroidal anti-inflammatory drugs and oral contraceptives, which may have adverse effects. Viburnum opulus (Cramp bark) is a homoeopathic remedy well indicated for the treatment of dysmenorrhea. While there are studies using Viburnum opulus in its herbal form, there is no research assessing its efficacy in the homoeopathic form.

The aim of this study is to determine the efficacy of Viburnum opulus 3X in the treatment of primary dysmenorrhea as measured with the modified Short Form McGill pain questionnaire (SF-MPQ-2) and visual analogue scale (VAS) respectively.

DETAILED DESCRIPTION:
This will be a double blind placebo controlled study, involving 30 female participants. The study will run for 3 months, over 3 menstrual cycles and shall be determined by the length of each participant menstrual cycle. The participants will be assessed over 3 menstrual events. Consultations will take place in a private setting at the Homoeopathic Health Centre at the Doornfontein campus, under the supervision of a registered homoeopath.

Participants will be recruited by advertisements placed at the University of Johannesburg Health Centre located on the Doornfontein campus, with the relevant permission obtained.

The researcher will explain the study to each participant as well as provide each participant with a consent form to sign, before they may take part in the study. Participants will be screened and a general physical examination will be conducted to asses each participant's general wellbeing. Each participant will be issued with a modified Short Form McGill questionnaire and the Visual Analogue Scale to complete. Participants will be instructed to complete the forms when they begin to experience the pain and cramping. No medication will be given at the initial consultation.

During the second follow-up consultation the participants will return their completed forms given to them at the initial consultation. Each participant will be issued with a 50 ml bottle of the homoeopathic remedy or placebo and new forms (SF-MPQ-2 and VAS) to complete. Participants will be advised to take 10 drops of the remedy three times a day starting when they experience pain and cramping. The forms will additionally need to be completed during this time. The participants will be advised to stop the homoeopathic remedy when their pain and cramping has ceased. This process will be repeated at both the third and fourth consultations.

During the final consultation participants will return the last forms to the researcher. The participants will measure their subjective satisfaction of the medicine on their pain by completing the five point treatment satisfaction scale.

The data will be statistically analysed by the researcher with the aid of a statistician. This will be done using the non-parametric Friedmann test (to measure the differences within both groups) and the Mann-Whitney test (to measure the differences between the groups) as well as the repeated measures ANOVA. These tests will evaluate the change of severity of symptoms over time.

The possible benefits for those participating in the study may include an improvement in their symptoms of primary dysmenorrhea. This study will contribute to the medical knowledge and efficacy of the clinical management of primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Females between 18-35 years.
* Have a history of painful menstruation.

Exclusion Criteria:

* Are on any form of hormonal contraceptives.
* Have intra uterine contraceptive devices.
* Have prediagnosed endometriosis, chronic pelvic inflammatory disease, uterine fibroids, polycystic ovarian syndrome or other known causes of secondary dysmenorrhea.
* Suffers from any serious chronic disease.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pain as measured by the Short Form McGill Pain Questionnaire (SF-MPQ-2) | 3 months
  The SF-MPQ-2 is a highly reliable and sensitive instrument used to asses and measure pain levels.

SECONDARY OUTCOMES:
Pain as measured by the Visual Analogue Scale (VAS) | 3 months
  The scale (VAS) is a validated and established tool used clinically to assess pain levels.
Patient satisfaction as measured by the 5-Point Treatment Satisfaction Scale | 1 day
  The 5-Point Treatment Satisfaction Scale is a reliable tool to assess patient satisfaction with the treatment provided. This will be conducted once at the final consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Solomon, D.TechHom, Study Director — University of Johannesburg
Locations (1):
- University of Johannesburg, Johannesburg, Gauteng, South Africa